CLINICAL TRIAL: NCT03125304
Title: Acupuncture for Pain of Endometriosis: A Multicenter, Randomized, and Controlled Trial
Brief Title: Acupuncture for Pain of Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State Administration of Traditional Chinese Medicine of the People's Republic of China (Other Government)
Collaborators: The Affiliated Hospital of JiangXi University of TCM (Unknown); The Qionghai Hospital of TCM (Unknown); The GanZhou Maternal and Child Health Hospital (Unknown); The Second Affiliated Hospital of JiangXi University TCM (Unknown)
Responsible Party: Principal Investigator, Liang Ruining, Professor, Jiangxi University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: jdzy2015065
Record Dates: First submitted 2017-04-17; First posted 2017-04-24 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Endometriosis
Keywords: Endometriosis; acupuncture; pain; dysmenorrhea
MeSH Terms: conditions — Endometriosis; Pain; Dysmenorrhea | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: The participants assigned to the treatment groups will receive acupuncture at Sanyinjiao (SP 6), Zhaohai (KI 6) ,Taichong (LR 3) ,Qichong (ST 30) and Guanyuan (CV4), while the control group will receive acupuncture at non-acupoint.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Treatment group will receive acupuncture at Sanyinjiao (SP 6), Zhaohai (KI 6) ,Taichong (LR 3) ,Qichong (ST 30) and Guanyuan.
  Interventions: Other: acupuncture
- control group (Placebo Comparator): Control group will receive acupuncture at non-acupoints.
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — They will be treated seven days before expected menstrual onset with once a day and three times a week for therapy. During the menstrual period,they will be treated everyday when they are having pain.Every treatment lasts 30 minutes. The trial period will consist of three menstrual cycles of treatment and three menstrual cycles in the follow-up period.

SUMMARY:
This proposed trial is a multicenter,randomized and controlled clinical trial. The aim of this trial is to evaluate the efficacy and safety of acupuncture for treating pain of Endometriosis.The trial period will consist of three menstrual cycles of treatment, and three menstrual cycles in the follow-up period.We put forward the following hypothesis: the effect of acupuncture group is better than the control group on relieving pain.

DETAILED DESCRIPTION:
Endometriosis is a kind of chronic gynaecology disease that endometrial tissue appear outside the uterine cavity , the main symptoms include dysmenorrhea, dyspareunia, chronic pelvic pain, and infertility, etc. .The secondary progressive and aggravating dysmenorrhea is thought to be the most typical symptom of endometriosis.The epidemiology data shows that about 87.7% endometriosis patients accompany with dysmenorrhea, affecting majority of women's physical and mental health and quality of life seriously .The treatment for dysmenorrhea is still the key and pressing problem of endometriosis.Endometriotic lesions can be excised or ablated surgically, but the risk of recurrence is high. Drug therapy mainly involves the use of oral contraceptives, progesterone and androgen derivatives, gonadotropin-releasing hormone (GnRH) agonists and aromatase inhibitors, etc.,However, in some women the side effects may not be well tolerated or the pain relief provided may be inadequate. Therefore, a large number of patients with endometriosis are turning to complementary and alternative medicine such as acupuncture.Acupuncture, as an important component of traditional Chinese medicine is widely used in Asian countries,and it can treat different diseases, including endometriosis dysmenorrhea.The analgesia principle of acupuncture is based on the theory of holistic view of zang-fu organs and meridians.In traditional Chinese medicine, dysmenorrhea is etiologically caused by the stagnated blood or Qi circulation in the uterus. The pathological factors are mostly dampness, blood stasis,and Qi obstructions. Acupuncture stimulation, which involves thrusting or twisting needles,results in various biochemical reactions that can have effects throughout the body.When the running of blood and Qi is unobstructed, pain can be relieved.However, only some small trials considered to be lacking in quality or size to guide practice.So it is urgently necessary to design multicenter ,randomized controlled trial to prove it .

ELIGIBILITY:
Inclusion criteria

1. Women age between 20 and 40.
2. Endometriosis diagnosed according to the Endometriosis Consensus Guidelines (Chinese Medical Association, 2015): 1) symptomatic endometriosis detected by laparoscopy or laparotomy; or 2) ovarian endometrioma detected by ultrasound or magnetic resonance imaging with pelvic pain.
3. Patients willing to receive acupuncture for pain relief.
4. Pelvic pain score equal or over 4 cm on the Visual Analogue Scale (VAS).
5. Regular menstrual cycle.
6. Signed informed consent

Exclusion criteria

1. Pelvic ultrasound demonstrates the endometrial cyst measures more than 5 cm in diameter and surgery is indicated.
2. Imaging examination suspects pelvic genital malignancies.
3. Cancer antigen-125 > 200 IU/L.
4. Pelvic infectious diseases.
5. Other severe disorders in heart, lung, liver, kidney, or mental disorders not able to cooperate in the study.
6. Patients who have received any other treatment for endometriosis that may affect the observation of the curative effects of acupuncture these three months.
7. Pregnancy or breastfeeding.
8. Refusal to be randomized.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 106 (Actual)
Dates: Start 2017-05-21 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | up to 24 weeks
  Pelvic pain

SECONDARY OUTCOMES:
Endometriosis Health Profile -30 | up to 24 weeks
  Endometriosis-specific quality of life
Multidimensional Pain Inventory | up to 24 weeks
  Physical functioning
Beck Depression Inventory and Profile of Mood States | up to 24 weeks
  Emotional functioning
Patient Global Impression of Change | up to 24 weeks
  Patient satisfaction
Pain diary | up to 24 weeks
  the specific time and frequency of pain attacks, the duration of pain

CONTACTS AND LOCATIONS:
Overall Officials: Ruining Liang, Study Director — The Second Affiliated Hospital of Jiangxi University of TCM
Locations (1):
- the second affiliated hospital of Jiangxi University of TCM, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xiang DF, Sun QZ, Liang XF. [Effect of abdominal acupuncture on pain of pelvic cavity in patients with endometriosis]. Zhongguo Zhen Jiu. 2011 Feb;31(2):113-6. Chinese. PMID 21442808
- [Background] Rubi-Klein K, Kucera-Sliutz E, Nissel H, Bijak M, Stockenhuber D, Fink M, Wolkenstein E. Is acupuncture in addition to conventional medicine effective as pain treatment for endometriosis? A randomised controlled cross-over trial. Eur J Obstet Gynecol Reprod Biol. 2010 Nov;153(1):90-3. doi: 10.1016/j.ejogrb.2010.06.023. Epub 2010 Aug 21. PMID 20728977
- [Background] Zhang X, Li W. [Efficacy on endometriosis treated with electroacupuncture]. Zhongguo Zhen Jiu. 2015 Apr;35(4):323-6. Chinese. PMID 26054137
- [Background] Magalhaes J. Acupuncture for pain in endometriosis. Sao Paulo Med J. 2013;131(6):439. doi: 10.1590/1516-3180.20131316T1. PMID 24346786
- [Derived] Li PS, Peng XM, Niu XX, Xu L, Hung Yu Ng E, Wang CC, Dai JF, Lu J, Liang RN. Efficacy of acupuncture for endometriosis-associated pain: a multicenter randomized single-blind placebo-controlled trial. Fertil Steril. 2023 May;119(5):815-823. doi: 10.1016/j.fertnstert.2023.01.034. Epub 2023 Jan 27. PMID 36716811
- [Derived] Liang R, Li P, Peng X, Xu L, Fan P, Peng J, Zhou X, Xiao C, Jiang M. Efficacy of acupuncture on pelvic pain in patients with endometriosis: study protocol for a randomized, single-blind, multi-center, placebo-controlled trial. Trials. 2018 Jun 7;19(1):314. doi: 10.1186/s13063-018-2684-6. PMID 29880009